CLINICAL TRIAL: NCT01420783
Title: A Randomized Phase II, Open-Label Study of the Efficacy and Safety of Orally Administered SAR302503 in Patients With Polycythemia Vera (PV) or Essential Thrombocythemia (ET) Who Are Resistant or Intolerant to Hydroxyurea
Brief Title: Study With SAR302503 in Patients With Polycythemia Vera or Essential Thrombocythemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARD12042; 2011-001847-58 (EudraCT Number); U1111-1121-4203 (Other: UTN)
Record Dates: First submitted 2011-08-11; First posted 2011-08-22 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2016-02

CONDITIONS: Hematopoietic Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — fedratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- SAR302503 100 mg (Experimental): once daily X 28 days
  Interventions: Drug: SAR302503
- SAR302503 200 mg (Experimental): once daily X 28 days
  Interventions: Drug: SAR302503
- SAR302503 400 mg (Experimental): once daily X 28 days
  Interventions: Drug: SAR302503
- SAR302503 600 mg (Experimental): once daily X 28 days
  Interventions: Drug: SAR302503

INTERVENTIONS:
Drug: SAR302503 — Pharmaceutical form:capsule
  Route of administration: oral

SUMMARY:
Primary Objective:

* Dose Ranging Phase: To evaluate the efficacy of daily oral doses of 100, 200, and 400 mg SAR302503 in patients with PV and ET who are resistant or intolerant to hydroxyurea (per European LeukemiaNet criteria) for :

  * Inducing absence of phlebotomy and a hematocrit below 45% for a minimum of 3 months in patients with polycythemia vera, and
  * Reduction of platelet count to ≤400 x 10x9/L for a minimum of 3 months in patients with essential thrombocythemia.
* PV Dose Expansion Phase and ET Dose Ranging Phase (only 600 mg dose group): To evaluate the efficacy of daily oral SAR302503 in patients with PV and ET who are resistant or intolerant to hydroxyurea (per European LeukemiaNet criteria) for:

  * Inducing absence of phlebotomy eligibility beginning at Day 1 of Cycle 4 visit and continuing through Day 1 of Cycle 6 visit in patients with PV, and
  * Reduction of platelet count to ≤400 x 10x9/L beginning at Day 1 of Cycle 4 visit and continuing through Day 1 of Cycle 6 visit in patients with ET.

Secondary Objectives:

* To evaluate the safety of SAR302503.
* To evaluate the efficacy of SAR302503 in patients with PV who are resistant or intolerant to hydroxyurea for inducing absence of phlebotomy eligibility.
* To evaluate the efficacy of SAR302503 in patients with ET who are resistant or intolerant to hydroxyurea for reduction of platelet counts.
* To evaluate the efficacy of SAR302503 in inducing complete and partial responses beginning at Day 1 of Cycle 6 visit through Cycle 8.
* To evaluate splenic response as measured by spleen volume using MRI or CT.
* To evaluate the pharmacokinetics of SAR302503 after single and repeat doses.
* To evaluate the pharmacodynamics of SAR302503 as measured by changes in JAK2V617F allele burden in patients with JAK2V617F mutation, and STAT3 phosphorylation inhibition.
* To measure improvement in baseline myeloproliferative neoplasm (MPN)-associated symptoms, as well as overall impact on quality of life.
* To measure generic health-related quality of life and utility value using the EuroQol Group (EQ-5DTM) questionnaire.

DETAILED DESCRIPTION:
The duration of the study for an individual patient is at least 40 weeks and will include a period to assess eligibility (screening period) of up to 4 weeks (28 days), a treatment period of up to 8, 28-day cycles (32 weeks), and a follow-up visit 30 days following the last administration of study drug. Treatment may continue if the patient is deriving benefit and does not experience disease progression, unacceptable toxicity, or meet other study withdrawal criteria.

Per Protocol Amendment No. 5, accrual of patients with essential thrombocythemia is closed.

ELIGIBILITY:
Inclusion criteria:

* Has had a diagnosis of hydroxyurea resistant or intolerant polycythemia vera (PV) or essential thrombocythemia (ET) documented at Screening.
* Polycythemia vera or essential thrombocythemia defined according to the revised WHO criteria.
* Polycythemia vera resistance or intolerance to hydroxyurea is defined as polycythemia vera patients on hydroxyurea with a hematocrit >45%, or phlebotomy twice in the last 6 months and at least once in the last 3 months.
* Essential thrombocythemia resistance or intolerance to hydroxurea is defined as essential thrombocythemia patients on HU with platelet count >600 x 10x9/L.

Dose Expansion Phase (polycythemia vera) and 600 mg/day group (essential thrombocythemia):

* Has had a diagnosis of polycythemia vera or essential thrombocythemia according to the revised WHO 2008 criteria.
* PV patients must be resistant or intolerant to hydroxyurea.
* ET patients must be resistant or intolerant to hydroxyurea.
* Provide written informed consent to participate.

Exclusion criteria:

* Less than 18 years of age.
* Participation in any study of an investigational agent (drug, biologic, device) within 30 days prior to initiation of study drug, unless during non-treatment phase. (Prior treatment with another JAK2 inhibitor is allowed.)
* Unwilling to comply with scheduled visits, treatment plans, laboratory assessments, and other study-related procedures.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 3 or 4 at study entry.
* Splenectomy.
* Active malignancy other than polycythemia vera or essential thrombocythemia, except adequately treated basal cell carcinoma and squamous cell carcinoma of the skin, cervical carcinoma in situ, or other malignancies that have been stable and off therapy for ≥5 years.
* Major surgery within 28 days or radiation within 3 months prior to initiation of study drug.
* Active acute infection requiring antibiotics.
* Known human immunodeficiency virus or acquired immunodeficiency syndrome-related illness.
* Uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4), angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass surgery, transient ischemic attack, or pulmonary embolism within 3 months prior to initiation of study drug.
* Any severe acute or chronic medical, neurological, or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, may interfere with the informed consent process and/or with compliance with the requirements of the study, or may interfere with interpretation of study results and, in the Investigator's opinion, would make the patient inappropriate for entry into this study.
* Inadequate organ function.
* Known active (acute or chronic) Hepatitis A, B, or C; and Hepatitis B and C carriers.
* Prior history of chronic liver disease (eg, chronic alcoholic liver disease, autoimmune hepatitis, sclerosing cholangitis, primary biliary cirrhosis, hemachromatosis, non-alcoholic steatohepatitis [NASH]).
* Concomitant treatment with or use of drugs or herbal agents known to be at least moderate inhibitors or inducers cytochrome P450 3A4 (CYP3A4).
* Presence of any gastric or other disorder that would inhibit absorption of oral medication.
* Known hypersensitivity to any excipients in the study drug formulation.
* Women of childbearing potential, unless using effective contraception while on study drug.
* Men who partner with a woman of childbearing potential, unless they agree to use effective contraception while on study drug.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2011-10; Primary Completion 2012-11 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Dose Ranging Phase: Proportion of PV patients with absence of phlebotomy and hematocrit below 45% and proportion of ET patients with a platelet count ≤ 400 x 10x9/L for a minimum of 3 months during the first 8 cycles of therapy. | 2 years
PV Dose Expansion Phase: Proportion of PV patients with absence of phlebotomy eligibility beginning at Day 1 of Cycle 4 visit and continuing through Day 1 of Cycle 6 visit. | 2 years
ET Dose Ranging Phase (only 600 mg dose group): Proportion of ET patients with a platelet count ≤400 x 10x9/L beginning at Day 1 of Cycle 4 visit and continuing through Day 1 of Cycle 6 visit. | 2 years

SECONDARY OUTCOMES:
Proportion of PV patients with absence of phlebotomy eligibility beginning at Day 1 of Cycle 4 visit through Cycle 8 (for PV dose expansion phase only). | 2 years
Proportion of ET patients with platelet count ≤400 x 10x9/L beginning at Day 1 of Cycle 4 visit and continuing through Cycle 8. | 2 years
Characterization of clinicohematologic response (CR, PR, and no Response) defined by European LeukemiaNet beginning at Day 1 of Cycle 6 visit through Cycle 8. | 2 years
Percent change in spleen volume (per Magnetic Resonance Imaging (MRI)) at the end of Cycles 4 and 8 or end of treatment (EOT) relative to baseline. | 2 years
Proportion of patients with a ≥ 35% reduction in spleen volume (per Magnetic Resonance Imaging (MRI)) at the end of Cycles 4 and 8 or end of treatment (EOT) relative to baseline. | 2 years
Number of participants who have changes in histological, cytogenetic, and molecular responses in bone marrow. | 2 years
Response (defined as either a 2-point improvement in or resolution of a symptom present at baseline) at the end of Cycles 1, 4, and 8 or end of treatment (EOT), as measured by the Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF). | 2 years
Cumulative Distribution Function of responses between treatment groups at the end of Cycles 1, 4, and 8 or EOT on the MPN-SAF. | 2 years
For each MPN-associated symptom present at baseline on the MPN-SAF, proportion of patients with resolution of that symptom at the end of Cycles 1, 4, and 8. | 2 years
To measure generic health-related quality of life and utility values using the EQ-5D questionnaire after completion of 8 cycles of therapy. | 2 years
Characterization of the safety profile of SAR302503, including the frequency, duration, and severity of adverse events graded using the National Cancer Institute (NCI) - CTCAE version 4.03, clinical laboratory parameters, ECG, and vital signs. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (35):
- United States (8):
  - Investigational Site Number 840008, Scottsdale, Arizona
  - Investigational Site Number 840004, La Jolla, California
  - Investigational Site Number 840005, Los Angeles, California
  - Investigational Site Number 840011, Palo Alto, California
  - Investigational Site Number 840010, Ann Arbor, Michigan
  - Investigational Site Number 840007, Rochester, Minnesota
  - Investigational Site Number 840003, St Louis, Missouri
  - Investigational Site Number 840001, Houston, Texas
- Australia (4):
  - Investigational Site Number 036001, Clayton
  - Investigational Site Number 036002, Kingswood
  - Investigational Site Number 036004, Kogarah
  - Investigational Site Number 036003, Randwick
- Canada (3):
  - Investigational Site Number 124002, Montreal
  - Investigational Site Number 124003, Toronto
  - Investigational Site Number 124001, Vancouver
- France (3):
  - Investigational Site Number 250004, Brest
  - Investigational Site Number 250003, Marseille
  - Investigational Site Number 250001, Paris
- Germany (2):
  - Investigational Site Number 276004, Frankfurt am Main
  - Investigational Site Number 276003, Mannheim
- Italy (3):
  - Investigational Site Number 380003, Bologna
  - Investigational Site Number 380001, Florence
  - Investigational Site Number 380004, Orbassano
- South Korea (4):
  - Investigational Site Number 410001, Seongnam
  - Investigational Site Number 410003, Seoul
  - Investigational Site Number 410004, Seoul
  - Investigational Site Number 410002, Seoul
- Spain (4):
  - Investigational Site Number 724004, Badalona
  - Investigational Site Number 724001, Barcelona
  - Investigational Site Number 724003, Madrid
  - Investigational Site Number 724002, Valencia
- United Kingdom (4):
  - Investigational Site Number 826001, Belfast
  - Investigational Site Number 826006, Birmingham
  - Investigational Site Number 826003, London
  - Investigational Site Number 826004, London